CLINICAL TRIAL: NCT00435669
Title: Mass Balance, Pharmacokinetics and Metabolism of [14C]BMS-582664 Prodrug of BMS-540215, in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: A Phase I Study to Determine Absorption, Distribution, Metabolism, and Elimination of a Single Radiolabeled Dose of Brivanib (BMS-582664)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA182-008
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2008-07

CONDITIONS: Tumors
Keywords: Advanced or metastatic solid tumors
MeSH Terms: conditions — Neoplasms | interventions — brivanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Brivanib — Oral Solution, Oral, 800 mg, X1 on Day 1, 10 D for ADME
  Other Names: BMS-582664
Drug: Brivanib — Tablet, Oral, Brivanib 800 mg, QD, until progression

SUMMARY:
The purpose of this trial is to determine the mass balance, pharmacokinetics, metabolism, and routes and extent of elimination of BMS-582664

ELIGIBILITY:
Inclusion Criteria:

* Histologic/cytologic diagnosis of advanced or metastatic solid tumors
* ECOG 0-2
* 4/6 weeks since prior therapy

Exclusion Criteria:

* Brain metastases
* Secondary primary malignancy
* Thromboembolic disease requiring full anticoagulation within 6 months
* Inability to swallow or absorb oral therapy
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Absorption | Determined by PK measurement collected on Day 1 at timepoints 0 (predose) 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18 and 24 hour. Continue daily PK collection on Day 2 to Day 10
Distribution | Determined by PK measurement collected on Day 1 at timepoints 0 (predose) 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18 and 24 hour. Continue daily PK collection on Day 2 to Day 10
Metabolism | Determined by PK measurement collected on Day 1 at timepoints 0 (predose) 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18 and 24 hour. Continue daily PK collection on Day 2 to Day 10
Elimination of BMS-582664 | Determined by PK measurement collected on Day 1 at timepoints 0 (predose) 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18 and 24 hour. Continue daily PK collection on Day 2 to Day 10

SECONDARY OUTCOMES:
To assess safety and tolerability of BMS-582664 800 mg administered daily in Part B | at last patient last visit

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States